CLINICAL TRIAL: NCT02695355
Title: Pediatric Attention Deficit Hyperactivity Disorder: Predicting Clinical Response to Stimulant Medication From Single-dose Changes in Event Related Potentials
Brief Title: ERP Based Single-dose Predictions of Stimulants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB3330
Record Dates: First submitted 2016-02-15; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADHD medication effects (Experimental): Single dose methylphenidate (Ritalin tablets); 10 mg for ages 8-13; 15 mg for ages 13-17
  Interventions: Drug: Methylphenidate (MPH)

INTERVENTIONS:
Drug: Methylphenidate (MPH) — Test 1: No medication. Registration of ERPs and behavioral data during an attention task. Test 2: Test repeated on a single dose of MPH. Outcome measure: Classification as responders or non-responders after a four weeks medication trial, based on rating scales from parents and Teachers.
  Other Names: Ritalin tablets

SUMMARY:
The purpose of this study was to see if the clinical outcome of stimulant medication (methylphenidate) in pediatric Attention Deficit Hyperactivity Disorder can be predicted on the bases of changes in Event Related Potentials (ERPs) induced by a single dose of stimulant medication. (ERPs are extracted from electroencephalographic (EEG) registrations during the performance of an attention task).

DETAILED DESCRIPTION:
In the pediatric neuropsychiatric clinic of Ostfold Hospital Trust, Norway, patients diagnosed with attention deficit hyperactivity disorder are tested with quantitative EEG (QEEG) and ERPs to supplement the neuropsychological examination. In the majority of cases a systematic four weeks trial on stimulant medication is offered, and the clinical effects are evaluated at the end of the try-out period. This procedure is a clinical routine. In this study patients and parents were asked if they were willing to complete a second QEEG/ERP test on a single dose of stimulant medication shortly before the onset of the four weeks trial. They were explained that the aim of the study was to search for predictors of clinical response. They were also informed that this second test was completely voluntary. (In fact the vast majority were quite enthusiastic). The patients were characterized as responders (REs - medication continued) or non-responders (non-REs - medication stopped) based on explicit criteria. The single-dose induced changes in ERPs (and behavioral parameters from the attention test; number of errors, reaction times) were examined, and differences between REs and non-REs were calculated.

If the analysis of data show that one or several variables are significantly different in REs and non-REs with large effect sizes, these findings may eventually result in the development of a useful clinical tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the clinic diagnosed with Attention Deficit Hyperactivity Disorder. Cases With comorbid diagnoses such as emotional or behavioral disorders, learning disabilities or high functioning autism are included.

Exclusion Criteria:

* Patients With intelligence coefficients below 70 or a diagnosed neurological disease are excluded.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2006-10; Primary Completion 2013-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Classification as responders (REs) or non-responders (non-REs) based on daily ratings from parents and teachers of ADHD symptoms during a four weeks medication trial | Classification as RE or non-RE within a time frame of five to ten weeks after onset of medication trial.

CONTACTS AND LOCATIONS:
Overall Officials: Geir Ogrim, PhD, Principal Investigator — Ostfold Hospital Trust
Locations (1):
- Pediatric Neuropsychiatric Team, Østfold Hospital Trust, Fredrikstad, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ogrim G, Hestad KA, Brunner JF, Kropotov J. Predicting acute side effects of stimulant medication in pediatric attention deficit/hyperactivity disorder: data from quantitative electroencephalography, event-related potentials, and a continuous-performance test. Neuropsychiatr Dis Treat. 2013;9:1301-9. doi: 10.2147/NDT.S49611. Epub 2013 Sep 5. PMID 24043939
- [Result] Ogrim G, Kropotov J, Brunner JF, Candrian G, Sandvik L, Hestad KA. Predicting the clinical outcome of stimulant medication in pediatric attention-deficit/hyperactivity disorder: data from quantitative electroencephalography, event-related potentials, and a go/no-go test. Neuropsychiatr Dis Treat. 2014 Feb 3;10:231-42. doi: 10.2147/NDT.S56600. eCollection 2014. PMID 24523588
- [Result] Hermens DF, Cooper NJ, Kohn M, Clarke S, Gordon E. Predicting stimulant medication response in ADHD: evidence from an integrated profile of neuropsychological, psychophysiological and clinical factors. J Integr Neurosci. 2005 Mar;4(1):107-21. doi: 10.1142/s0219635205000653. PMID 16041867
- [Result] Johnston BA, Coghill D, Matthews K, Steele JD. Predicting methylphenidate response in attention deficit hyperactivity disorder: a preliminary study. J Psychopharmacol. 2015 Jan;29(1):24-30. doi: 10.1177/0269881114548438. Epub 2014 Sep 18. PMID 25237119
- [Result] Barkley RA. Predicting the response of hyperkinetic children to stimulant drugs: a review. J Abnorm Child Psychol. 1976;4(4):327-48. doi: 10.1007/BF00922531. PMID 794087
- [Result] Chabot RJ, Orgill AA, Crawford G, Harris MJ, Serfontein G. Behavioral and electrophysiologic predictors of treatment response to stimulants in children with attention disorders. J Child Neurol. 1999 Jun;14(6):343-51. doi: 10.1177/088307389901400601. PMID 10385840
- [Result] Riccio CA, Waldrop JJ, Reynolds CR, Lowe P. Effects of stimulants on the continuous performance test (CPT): implications for CPT use and interpretation. J Neuropsychiatry Clin Neurosci. 2001 Summer;13(3):326-35. doi: 10.1176/jnp.13.3.326. PMID 11514638
- [Result] Sangal RB, Sangal JM. Attention-deficit/hyperactivity disorder: use of cognitive evoked potential (P300) to predict treatment response. Clin Neurophysiol. 2006 Sep;117(9):1996-2006. doi: 10.1016/j.clinph.2006.06.004. Epub 2006 Aug 4. PMID 16890481
- [Result] Young ES, Perros P, Price GW, Sadler T. Acute challenge ERP as a prognostic of stimulant therapy outcome in attention-deficit hyperactivity disorder. Biol Psychiatry. 1995 Jan 1;37(1):25-33. doi: 10.1016/0006-3223(94)00075-E. PMID 7893855
- [Result] Czerniak SM, Sikoglu EM, King JA, Kennedy DN, Mick E, Frazier J, Moore CM. Areas of the brain modulated by single-dose methylphenidate treatment in youth with ADHD during task-based fMRI: a systematic review. Harv Rev Psychiatry. 2013 May-Jun;21(3):151-62. doi: 10.1097/HRP.0b013e318293749e. PMID 23660970
- [Result] Linssen AM, Vuurman EF, Sambeth A, Nave S, Spooren W, Vargas G, Santarelli L, Riedel WJ. Contingent negative variation as a dopaminergic biomarker: evidence from dose-related effects of methylphenidate. Psychopharmacology (Berl). 2011 Dec;218(3):533-42. doi: 10.1007/s00213-011-2345-x. Epub 2011 May 20. PMID 21597989
- [Derived] Ogrim G, Kropotov JD. Predicting Clinical Gains and Side Effects of Stimulant Medication in Pediatric Attention-Deficit/Hyperactivity Disorder by Combining Measures From qEEG and ERPs in a Cued GO/NOGO Task. Clin EEG Neurosci. 2019 Jan;50(1):34-43. doi: 10.1177/1550059418782328. Epub 2018 Jun 25. PMID 29940782
- [Derived] Aasen IE, Ogrim G, Kropotov J, Brunner JF. Methylphenidate selectively modulates one sub-component of the no-go P3 in pediatric ADHD medication responders. Biol Psychol. 2018 Apr;134:30-38. doi: 10.1016/j.biopsycho.2018.02.011. Epub 2018 Feb 21. PMID 29476840